CLINICAL TRIAL: NCT01242475
Title: A Phase IIa Specificity Trial of the Diagnostic Agent C-Tb, When Given Intradermally by the Mantoux Technique to Healthy Volunteers Previously Vaccinated With BCG
Brief Title: A Trial of the C-Tb Skin Test, When Given Intradermally to Healthy Volunteers Previously Vaccinated With BCG
Acronym: TESEC-03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: TESEC-03; 2009-017296-17 (EudraCT Number)
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Tuberculosis
Keywords: tuberculosis; rdESAT-6; CFP-10; skin test; diagnostic test
MeSH Terms: conditions — Tuberculosis | interventions — Tuberculin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.1µg/0.1 mL C-Tb (Experimental): The C-Tb and 2 TU Tuberculin PPD RT 23 SSI agents are given concomitantly to each volunteer in the RIGHT AND LEFT forearms according to a double blind randomisation scheme
  Interventions: Biological: C-Tb
- 2TU Tuberculin PPD RT 23 SSI (Active Comparator): The C-Tb and 2 TU Tuberculin PPD RT 23 SSI agents are given concomitantly to each volunteer in the RIGHT AND LEFT forearms according to a double blind randomisation scheme
  Interventions: Biological: 2 TU Tuberculin PPD RT 23 SSI

INTERVENTIONS:
Biological: C-Tb — The C-Tb agent is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearms according to a double blind randomisation scheme
  Other Names: rdESAT-6 + rCFP-10
  Arms: 0.1µg/0.1 mL C-Tb
Biological: 2 TU Tuberculin PPD RT 23 SSI — The 2TU Tuberculin PPD RT 23 SSI agent is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearms according to a double blind randomisation scheme
  Other Names: PPD; Tuberculin
  Arms: 2TU Tuberculin PPD RT 23 SSI

SUMMARY:
A new, more specific skin test to detect tuberculosis has been developed by Statens Serum Institut in Denmark. The new skin test is named C-Tb and like the current Tuberculin a positive test result will show as redness and/or swelling at the injection site, while a negative test will leave no reactions.

The aim of this study is to test the C-Tb skin test in healthy adults previously BCG vaccinated to determine if healthy non tuberculosis infected individuals has a truly negative test result (this is called determining the specificity of the skin test). To be able to compare the new skin test with the current Tuberculin skin test volunteers will be injected with both the C-Tb and the TST skin test.

DETAILED DESCRIPTION:
The trial is designed to investigate the specificity of C-Tb under various definitions of cut-off in a double blind randomised, split-body study comparing 0.1 µg/0.1 mL C-Tb with the reference agent 2 T.U. Tuberculin PPD RT23 SSI. (Each volunteer receives the C-Tb agent in one arm and the 2 T.U. Tuberculin PPD in the other arm).

The C-Tb and 2 T.U. Tuberculin PPD agents are given concomitantly to each volunteer in the RIGHT AND LEFT forearm according to a double blind randomisation scheme.

The primary objective of the trial is to assess the specificity of the C-Tb test as a function of the cut-off value (i.e., the smallest size of induration measured in mm resulting in a negative outcome of the C-Tb test) when the test is administered intradermally by the Mantoux technique to healthy BCG vaccinated adults The specificity of the C-Tb test is defined as the relative frequency of subjects in a healthy population (i.e., no exposure to MTb) who have an induration response < cut-off after a C-Tb test.

Similarly the sensitivity is defined as the relative frequency of patients with an induration response ≥ cut-off in TB patients.

An optimal cut-off point of being infected will be determined by combing the results from the present specificity study with those from a parallel sensitivity study in patients recently diagnosed with TB.

The secondary objectives of the trial are to compare the induration response of C-Tb with the induration response of 2 T.U. Tuberculin PPD RT 23 SSI, to compare the induration response of C-Tb with the in-vitro IFN-γ response measured at screening and 28 days after the injections of the skin test agents using the QuantiFERON®-TB Gold In-Tube assay and finally to record all adverse events occurring within 28 days after application of the agents.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed an informed consent
2. Aged 18 to 65 years
3. Is known to be BCG vaccinated (documented in medical files and/or by the presence of a BCG scar)
4. Is healthy according to a medical examination and medical history at screening
5. Is willing and likely to comply with the trial procedures
6. Is prepared to grant authorized persons access to their medical records

Exclusion Criteria:

1. Has a history of tuberculosis or has been in close contact to a person with active tuberculosis within 5 years from trial inclusion
2. Has a positive QuantiFERON®-TB Gold In-Tube assay at inclusion
3. Laboratory parameters outside of normal range judged by site investigator to be clinically significant
4. Has within 3 months prior to the day of inclusion been in treatment with a product which is likely to modify the immune response (e.g., immunoglobulin, systemic corticosteroids, methotrexate, azathioprine, cyclosporine or blood products)
5. Has been vaccinated with a live vaccine within 6 weeks prior to the day of inclusion (e.g. MMR, yellow fever, oral typhoid vaccines)
6. Has been vaccinated with BCG < 6 months prior to the day of inclusion
7. Has been tuberculin (TST) tested < 6 months prior to the day of inclusion
8. Has a known congenital or acquired immune deficiency
9. Has an active disease affecting the lymphoid organs (e.g., Hodgkin's disease, lymphoma, leukaemia, sarcoidosis)
10. Is infected with HIV
11. Has a current skin condition which interferes with the reading of the skin tests e.g. tattoos, severe scarring, burns/sunburns, rash, eczema, psoriasis, or any other skin disease at or near the injection sites
12. Has a condition where blood drawings pose more than minimal risk for the volunteer, such as haemophilia, other coagulation disorders, or significantly impaired venous access
13. Currently participating in another clinical trial with an investigational or non investigational drug or device, or has participated in another clinical trial within the 3 months prior to dosing
14. Has participated in previous clinical trials investigating the ESAT-6 and/or CPP-10 antigens
15. Is pregnant, breast-feeding or intending to get pregnant
16. Is a female not willing to use effective barrier (including spermicidal gel), hormonal or intrauterine contraceptive measures
17. Has a history of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence within the 12 months preceding Visit 1
18. Has a positive urine drug screen at Visit 1 and Visit 2 (i.e., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, or opiates)
19. Has a positive alcohol breath test at Visit 1 and Visit 2. [NOTE: subjects must be told to avoid consumption of alcoholic beverages for at least 24 hours prior to attending the Centre]
20. Has a condition which in the opinion of the investigator is not suitable for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The diameter of induration at the injection sites measured transversely to the long axis of the forearm 2-3 days after application of the agents | From injections to 2-3 days after application of the agents

SECONDARY OUTCOMES:
Injection site adverse reactions within 28 days after application of the agents | Onset between the injections and 28 days after the injections
All adverse events occurring within 28 days after application of the agents | Onset between the injections and 28 days after the injections
Laboratory safety parameters of haematology and biochemistry | Onset between the injections and 28 days after the injections
In vitro IFN-γ response as measured by the QuantiFERON®-TB Gold In-Tube assay from blood samples taken at screening and 28 days after the injections of the skin test agents | Onset between the injections and 28 days after the injections

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Thierry-Carstensen, Study Director — Statens Serum Institut; David JM Lewis, MD, Principal Investigator — Surrey Clinical Research Centre, University of Surrey
Locations (1):
- Surrey Clinical Research Centre, University of Surrey, Surrey, Guildford, Surrey, United Kingdom